CLINICAL TRIAL: NCT01702675
Title: Phase I, Monocentric, Double-blind, Randomized Study to Assess Tolerability, Safety and Pharmacokinetics of ACH15 After Single Dose and Multiple Doses in Healthy Male Volunteers
Brief Title: Study to Assess Tolerability, Safety and Pharmacokinetics of a New Drug
Acronym: ACH15
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ACH-HML-01(03/12)
Record Dates: First submitted 2012-09-26; First posted 2012-10-08 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Safety; Pharmacokinetics; Tolerability; Healthy men

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- ACH15 - 50mg capsule (Experimental): ACH15 50mg capsule by mouth single dose (Group 1)
  Interventions: Drug: ACH15 50 mg
- ACH15 - 250 mg capsule (Experimental): ACH15 250mg capsule by mouth as single dose(Group 2)
  Interventions: Drug: ACH15 250 mg
- ACH15 - 500mg capsule (Experimental): ACH15 500mg capsule by mouth in a single dose(Group 3)
  Interventions: Drug: ACH15 500mg
- ACH15 - 1000 mg (two 500mg capsule) (Experimental): ACH15 500mg capsule by mouth, two 500 mg capsules once as a single dose(Group 4)
  Interventions: Drug: ACH15 - 1000mg
- ACH15 - 2000 mg (four 500 mg capsule) (Experimental): ACH15 500mg capsule by mouth, four 500 mg capsules once as a single dose(Group 5)
  Interventions: Drug: ACH15 - 2000mg
- ACH15 - 500 mg (twice a day for 7 days) (Experimental): ACH15 500mg capsule by mouth twice a day for seven days (Group 6)
  Interventions: Drug: ACH15 - 500mg
- Placebo - 250 mg capsule (Placebo Comparator): Placebo 250mg capsule by mouth single dose (Group 2)
  Interventions: Drug: Placebo 250 mg
- Placebo - 500 mg capsule (Placebo Comparator): Placebo 500mg capsule by mouth in a single dose(Group 3)
  Interventions: Drug: Placebo 500mg
- Placebo - 1000 mg (two 500mg capsule) (Placebo Comparator): Placebo 500mg capsule by mouth, two 500 mg capsules once as a single dose(Group 4)
  Interventions: Drug: Placebo 1000mg
- Placebo 2000 mg (four 500mg capsule) (Placebo Comparator): Placebo 500mg capsule by mouth, four 500 mg capsules once as a single dose(Group 5)
  Interventions: Drug: Placebo 2000mg
- Placebo - 500 mg (twice a day for 7 days) (Placebo Comparator): Placebo 500mg capsule by mouth twice a day for seven days (Group 7)
  Interventions: Drug: Placebo 500mg

INTERVENTIONS:
Drug: ACH15 50 mg — ACH15 50mg capsule
  Arms: ACH15 - 50mg capsule
Drug: ACH15 250 mg — ACH15 250mg capsule
  Arms: ACH15 - 250 mg capsule
Drug: ACH15 500mg — ACH15 500 mg capsule
  Arms: ACH15 - 500mg capsule
Drug: ACH15 - 1000mg — ACH15 500mg capsule - two 500mg capsules in single dose
  Arms: ACH15 - 1000 mg (two 500mg capsule)
Drug: ACH15 - 2000mg — ACH15 500mg capsule (four 500mg capsules in one dose)
  Arms: ACH15 - 2000 mg (four 500 mg capsule)
Drug: ACH15 - 500mg — ACH15 - 500mg twice a day for 7 days
  Arms: ACH15 - 500 mg (twice a day for 7 days)
Drug: Placebo 250 mg — Capsule manufactured to mimic ACH15 250 mg capsule
  Arms: Placebo - 250 mg capsule
Drug: Placebo 500mg — Capsule manufactured to mimic ACH15 500 mg capsule
  Arms: Placebo - 500 mg (twice a day for 7 days); Placebo - 500 mg capsule
Drug: Placebo 1000mg — Capsule manufactured to mimic ACH15 500 mg capsule Placebo 500mg (two 500 mg capsules in one dose)
  Arms: Placebo - 1000 mg (two 500mg capsule)
Drug: Placebo 2000mg — Capsule manufactured to mimic ACH15 500 mg capsule Placebo 500mg (four 500 mg capsules in one dose)
  Arms: Placebo 2000 mg (four 500mg capsule)
Drug: Placebo 500mg — Capsule manufactured to mimic ACH15 500 mg capsule Placebo 500mg (500 mg capsules twice a day for 7 days)
  Arms: Placebo - 500 mg (twice a day for 7 days); Placebo - 500 mg capsule

SUMMARY:
The purpose of this study is evaluate the safety and tolerability parameters regarding the new drug in healthy men and evaluate the pharmacokinetics parameters after one dose and multiple doses of the new drug.

ELIGIBILITY:
Inclusion Criteria:

* Male patient, aged between 18 and 50 years;
* Body weight ≥ 50 kg and BMI ≥ 18.5 kg/m2 and ≤ 30 kg/m2;
* Healthy men accordance with their historical and tests;
* Healthy subject with laboratory results within the normal range or within the parameters accepted by the clinical protocol
* Negative results for parasitological stool examination performed in the clinical study;
* Subject of research with laboratory results within the normal range for urinalysis collected before the first visit;
* Research subjects allocated in Group 6 with endoscopy within the normal range;

Exclusion Criteria:

* History of gastrointestinal disease, hepatic, renal, cardiovascular, pulmonary, neurologic, hematologic, diabetes or glaucoma;
* Evidence on clinical examination or physical or complement, organ dysfunction or any clinically significant deviation from normality;
* History of use of psychotropic drugs or excessive alcohol consumption (more than two units of alcohol per day, one unit being equivalent to one cup (200 mL) of brew or a dose (50) mL of distilled beverage) or having difficulty to abstain during the study;
* Use of any medication two (2) weeks prior to inclusion of the research subject in the study;
* Regular smokers or who quit less than one (1) year;
* History of food allergy or hyperreactivity to medications or foods;
* HIV positive for HIV;
* Being positive for Hepatitis B;
* Being positive for hepatitis C;
* Testing positive for Helicobacter pilorum;
* Using substances modulating hepatic microsomal activity within thirty (30) days prior to entry of the subject of research in the clinical study (date of signing the consent form);
* Having donated blood (blood volume higher than 500 mL) within four (4) months preceding the date of signing the consent form;
* Subject with a history of hypersensitivity to any component of the investigational product;

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 30 days
Electrocardiogram | 30 days
Echocardiography (participants included in Group 6) | 30 days
Cmax | 31 time points up to 2 days
  Blood analysis to evaluate drug pharmacokinetics at Group 1 to 5: 30 minutes and 05 minutes before dose and 00h10 min, 00h15 min, 00h30 min, 00h45 min, 01h, 01h15min, 01h30min, 01h45min, 02h, 02h15min, 02h30min, 02h45min, 03h, 03h15min, 03h30min, 03h45min, 04 h, 04h15min, 04h30min, 04h45min, 05h, 05h30min, 06 h, 08 h, 10 h, 12h, 16h, 24 h e 48hours post-dose
High digestive endoscopy (participants included at Group 6) | 8 days
  Image exam to evaluate the drug safety
Blood analysis | 30 days
  Blood will be collected to evaluate the drug safety by analysis of biochemical profile
Cmax | 67 pint time over 8 days
  Blood analysis to evaluate drug pharmacokinetics at Group 6:00:30 min before dose, 00h20min, 00h40min, 01h, 01h15min, 01h30min, 01h45min, 02h, 02h15min, 02h30min, 02h45min, 03h, 03h15min, 03h30min, 03h45min, 04h, 04h15min, 04h30min, 04h45min, 05h, 05h30min, 06h, 08h, 10h, 12h, 14h, 18h, 24h, 26h, 30h, 36h, 38h, 42h, 48h, 50h, 54h, 60h, 62h, 66h, 72h, 74h, 78h, 84h, 86h, 90h, 96h, 98h, 102h, 108h, 110h, 114h, 120h, 122h, 126h, 132h, 134h, 138h, 144h, 146h, 150h, 156h, 158h, 162h, 168h, 174h, 180h e 192h post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Vencio, MD, Principal Investigator — ICF - Instituto de Ciências Farmacêuticas
Locations (1):
- ICF - Instituto de Ciências Farmacêuticas, Aparecida de Goiânia, Goiás, Brazil